CLINICAL TRIAL: NCT06348173
Title: Response and Remission to Treatment With Anti-IL5/IL5R Antagonists in a Real-world Setting
Brief Title: Response and Remission to Treatment With Anti-IL5/IL5R Antagonists
Status: Completed | Type: Observational
Sponsor: Université de Montréal (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-2190
Record Dates: First submitted 2024-03-28; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — mepolizumab; benralizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Mepolizumab — Compare the response to mepolizumab and benralizumab before and after treatment
  Other Names: benralizumab

SUMMARY:
The aim of this retrospective observational study is to compare the response and remission rate after treatment with IL5/IL5-R antagonists in asthmatics who would and would have not met the inclusion criteria of the original randomized clinical trials.

This study will be performed using the charts of the patients.

DETAILED DESCRIPTION:
Objective To compare the response and remission rate after treatment with IL5/IL5-R antagonists in asthmatics who would and would have not met the inclusion criteria of the original RCTs.

After having obtained authorization from the ethics committee of the CIUSSS du nord de l'île de Montréal and from the director of the Professional Services, all the charts of patients who received anti IL5/IL-5R at the tertiary asthma clinic of the Hôpital du Sacré-Coeur de Montréal will be reviewed.

Patients aged 75 years or younger, with a smoking history of less than 10 pack-year, and a FEV1 <80% predicted with reversibility in the previous year will be considered to fulfill the RCTs criteria. Response to treatment was defined by at least a 50% reduction in asthma exacerbations or in oral corticosteroids (OCS) doses in the year following the initiation of IL5/IL5R antagonists. Clinical remission on treatment at one year was defined as no exacerbation, no OCS and la 10% or less decrease in pre-bronchodilator FEV1 compared with baseline value.

ELIGIBILITY:
Inclusion Criteria:

Patients 18 years and older who were followed at the outpatient asthma clinic of Sacre-Cœur Hospital and have been treated with anti-IL5/il5R between 2016 and 2020.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients 18 years and older who were followed at the outpatient asthma clinic of Sacre-Cœur Hospital and have been treated with anti-IL5/il5R between 2016 and 2020.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Response to IL5/IL5R antagonists one year after cohort entry among subjects fulfilling and not fulfilling the original RCT inclusion criteria | one year
  A response to treatment was defined as a reduction of asthma exacerbations of at least 50% or a 50% or higher reduction of the OCS doses for steroid dependant patients in the year following the initiation of an IL5/IL5R antagonist compared to the year preceding the initiation of the treatment.
Remission rate with IL5/IL5R antagonists one year after cohort entry in subjects fulfilling and not fulfilling the original RCT inclusion criteria | One year
  Clinical remission on treatment at one year post cohort entry was defined as no asthma exacerbation, no treatment with OCS and a 10% or less decrease in pre-bronchodilator FEV1 compared with baseline value.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Lemiere, MD, Principal Investigator — Université de Montréal
Locations (1):
- Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No